CLINICAL TRIAL: NCT06133764
Title: Analysis of Odontogenic Keratocyst Treated With Various Modalities Over a 10-year
Brief Title: Risk-Adapted Treatment Strategies for Odontogenic Keratocysts: A Long-Term Randomized Clinical Trial Quantifying Recurrence Reduction
Acronym: OKCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ghada Amin Khalifa, PhD, Professor of Maxillofacial Surgery and Diagnostic Science, Qassim University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-40-03
Record Dates: First submitted 2023-11-08; First posted 2023-11-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Odontogenic Cysts
Keywords: Odontogenic cysts; Odontogenic Keratocysts
MeSH Terms: conditions — Odontogenic Cysts | interventions — Decompression; Eudragit E PO

STUDY DESIGN:
Intervention Model Description: The patents will be divided into five groups according to the treatment modalities used to treat their odontogenic cysts
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients, investigators, and outcomes assessor will not be informed about the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Enucleation + Peripheral ostectomy + Carnoy's solution chemical cauterization (E+ PO+ CS) (Experimental): The odontogenic keratocysts will be treated using enucleation, followed by peripheral ostectomy and then Carnoy's solution
  Interventions: Procedure: Enucleation+ Peripheral Ostectomy+Carnoy's solution chemical cauterization (E+CS + PO)
- Decompression/marsupialization (D/M) (Experimental): The odontogenic keratocysts will be managed by either Decompression or marsupialization
  Interventions: Procedure: Decompression/ marsupialization (D/M)
- Enucleation (E) (Experimental): The odontogenic keratocysts will only be managed by Enucleation (E)
  Interventions: Procedure: Enucleation (E)
- Enucleation+Carnoy's solution (E+CS) (Experimental): odontogenic keratocysts will be managed by Enucleation, followed by Carnoy's solution
  Interventions: Procedure: Enucleation+Carnoy's solution (E+CS)
- Enucleation+ Peripheral Ostectomy (E+PO) (Experimental): The odontogenic keratocysts will be treated using Enucleation, followed by peripheral ostectomy (E+PO)
  Interventions: Procedure: Enucleation+ Peripheral Ostectomy (E+ PO)

INTERVENTIONS:
Procedure: Enucleation+ Peripheral Ostectomy+Carnoy's solution chemical cauterization (E+CS + PO) — The enucleation procedures, which were meticulously carried out in order to remove the odontogenic keratocyst in one piece without breaking its lining or leaving any epithelial remnants.The peripheral ostectomy treatment will be carried out with a large spherical bur and plenty of irrigation.After filling the bone cavity with more sterile gauze, the Carnoy's solution was slowly injected into it with a plastic syringe. The gauze was continuously injected with CS until it was fully saturated without leaking too much into the surrounding tissues. The CS was held in place for 3 minutes.
  Other Names: (E + PO+ CS)
  Arms: Enucleation + Peripheral ostectomy + Carnoy's solution chemical cauterization (E+ PO+ CS)
Procedure: Decompression/ marsupialization (D/M) — A surgical window will be created in the cyst wall to drain the contents while retaining continuity between the cyst and the oral cavity
  Other Names: D/M
  Arms: Decompression/marsupialization (D/M)
Procedure: Enucleation (E) — The enucleation will be accomplished in the same manner that it will be performed in the group of Enucleation+ Peripheral Ostectomy+Carnoy's solution chemical cauterization (E+ PO+ CS).
  Other Names: E
  Arms: Enucleation (E)
Procedure: Enucleation+Carnoy's solution (E+CS) — Both enucleation and Carnoy's solution will be carried out as planned in the group Enucleation+ Peripheral Ostectomy+Carnoy's solution chemical cauterization (E+ PO+ CS).
  Other Names: (E+CS)
  Arms: Enucleation+Carnoy's solution (E+CS)
Procedure: Enucleation+ Peripheral Ostectomy (E+ PO) — Both enucleation and peripheral ostectomy will be carried out as planned in the group Enucleation+ Peripheral Ostectomy+ Carnoy's solution chemical cauterization (E+ PO+ CS).
  Other Names: (E+PO)
  Arms: Enucleation+ Peripheral Ostectomy (E+PO)

SUMMARY:
Background The odontogenic keratocysts (OKCs) have been one of the maxillofacial region's most contentious pathological phenomena. Decompression/marsupialization (D/M), enucleation (E), enucleation + chemical cauterization with Carnoy's solution (E+CS), enucleation + peripheral ostectomy (E + PO), as opposed to enucleation + chemical cauterization with Carnoy's solution + peripheral ostectomy (E + CS + PO), were used during surgery to ensure that no epithelial remnants were left behind.

Rationale Through the management of OKC a recurrence could occur, the effectiveness of Decompression/marsupialization (D/M), Enucleation (E), Enucleation+Carnoy's solution chemical cauterization (E+CS), Enucleation+peripheral ostectomy (E+PO), Enucleation+Carnoy's solution chemical cauterization + peripheral ostectomy (E+CS + PO), will be analyzed

DETAILED DESCRIPTION:
Since the middle of the 20th century, the odontogenic keratocyst (OKC) has been one of the maxillofacial region's most contentious pathological phenomena. It was initially misdiagnosed as a primordial cyst. After that, because of its severe clinical behavior and tendency to recur, it was no longer considered to be a part of its classification, also known as a odontogenic tumor. Then, In 2017, the OKC are re-classified as a cystic lesion. But still there is debate about their management. So, this study will be enrolled with the following objectives: to describe how odontogenic keratocysts are managed, to Discover the most favorable approach to manage OKC with the need to stop it from happening again To categorize the odontogenic keratocyst management outcomes into to the subsequent groups: (1) total resolution, (2) partial resolution; (3) Recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All odontogenic keratocysts that are treated by the following surgical treatment modalities:

  1. Enucleation followed by peripheral ostectomy and Carnoy's solution
  2. Decompression/ marsupialization
  3. Enucleation
  4. Enucleation and Carnoy's solution
  5. Enucleation and Peripheral Ostectomy
* Follow-up period 10 years

Exclusion Criteria:

* Cases treated with resection
* Cases showed neoplastic transformation in their pathology
* Cyst Like lesions

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Healing period | Starting from the postoperative third month up to the postoperative ninth month
  The bone filling will monitored by using computed tomography scans
Measurement of the bony cavity | At the end of the postoperative ninth month
  A presence of radiolucent area in the computed tomography scans
Recurrence rate | At the end of the postoperative fifth year
  The new occurrence of the previously removed odontogenic keratocyst will be documented
Recurrence rate | At the end of the postoperative tenth year
  The new occurrence of the previously removed odontogenic keratocyst will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Khalifa, Professor, Principal Investigator — College of Dentistry, Qassim University, Saudi Arabia
Locations (1):
- College of Dentistry, Qassim University, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All data will be available on request by contact the principle investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after publication
Access Criteria: Contact the principle investigator via email: g.khalifa@qu.edu.sa